CLINICAL TRIAL: NCT02491840
Title: Biomoleculars Markers of Sensitivity to Pre- and Post-operative Chemotherapy of Gastric and Cardia Adenocarcinomas: a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6042
Record Dates: First submitted 2015-06-23; First posted 2015-07-08 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Gastric and Cardia Adenocarcinomas
Keywords: gastric cancer; cardia cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gastric and cardia adenocarcinomas (Experimental): Biopsy of Gastric and cardia adenocarcinomas
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsy of Gastric and cardia adenocarcinomas

SUMMARY:
Some subtypes of gastric and cardia tumors such as adenocarcinoma or gastric linitis with disseminated cells respond poorly to the pre-operative chemotherapy, and some of them do not respond to chemotherapy usually performed. Doing chemotherapy in these patients could delay their surgical management. The completion of chemotherapy for these patients would be a bad prognosis factor according to recent data from the literature. Therefore, the aim of this research is to find prognostic markers of sensitivity to chemotherapy usually performed. The investigators are going to use biopsies realized at diagnosis and select patients "good and bad" responders.

Primary purpose:

To study cardia and gastric tumors, molecular markers sensitivity to pre- and post- perative chemotherapy protocols (EOX protocol ... FOLFOX) or chemoradiation

Secondary purposes:

* To assess the impact of patients' lifestyle (via a questionnaire) on the response to chemotherapy
* To study markers of cancer stem cells
* To correlate clinical and molecular markers with patient survival and quality of life questionnaires
* To characterize the expression levels (Met, Her2, FGFR2) and mutations (p53 ras) in frequently deregulated genes in gastric cancers.
* To characterize the level of expression of predictive candidate markers (ΔNp73, TAp73, HDAC4, mir140, EZH2, CXCL12, CXCR4, CXCR7) found in the literature.
* To correlate the abnormalities found in the with tumor stages (before and after chemotherapy) and with 5 years overall survival and progression-free patients

ELIGIBILITY:
Inclusion Criteria:

Gastric adenocarcinoma (any location) or cardia adenocarcinoma

* Age> 18 years
* WHO Index≤ 3
* Subject having signed an informed consent

Exclusion Criteria:

* Other cancers undergoing chemotherapy treatment
* Pregnant or breastfeeding
* Inability to understand information (understanding with difficulties ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of expression level of Met | at 15 days
  To search in gastric and cardia tumors molecular markers of sensitivity to pre- and post-operative chemotherapy protocols (EOX protocol ... FOLFOX) or chemoradiation
Assessment of expression level of Her2 | at 15 days
  To search in gastric and cardia tumors molecular markers of sensitivity to pre- and post-operative chemotherapy protocols (EOX protocol ... FOLFOX) or chemoradiation
Assessment of expression level of FGFR2 | at 15 days
  To search in gastric and cardia tumors molecular markers of sensitivity to pre- and post-operative chemotherapy protocols (EOX protocol ... FOLFOX) or chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Benoît ROMAIN, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France